CLINICAL TRIAL: NCT05592990
Title: A Two Part, Randomized, Participant and Investigator-blinded, 2-arm, Parallel-design, Placebo-controlled Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of NGI226 Microparticles on Tendon Regeneration in Patients With Achilles Tendinopathy
Brief Title: A Study to Investigate the Safety, Tolerability and Preliminary Efficacy of NGI226 Microparticles in Patients With Achilles Tendinopathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNGI226A12201; 2022-500863-10-00 (Other: EU CT)
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Achilles Tendinopathy
Keywords: Achilles tendon; mid-portion Achilles tendinopathy; peritendon injection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NGI226 (Experimental): single peritendon injection
  Interventions: Drug: NGI226
- Placebo (Placebo Comparator): single peritendon injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NGI226 — NGI226 MP
  Arms: NGI226
Drug: Placebo — Placebo MP
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure local and systemic safety and tolerability as well as improvement of Achilles tendon mechanical properties after a single peritendon injection of NGI226 MP in comparison to placebo MP in patients with mid-portion Achilles tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to all study specific screening procedures, as close to the start of the screening period as possible.
* Presence of clinically (local Achilles tendon pain on tendon-loading activities, pain on palpation at the level 2-6 cm proximal to the calcaneal insertion) and ultrasound (local tendon thickening with hypoechogenicities and irregular fibre orientation) or MRI diagnosed mid-portion Achilles tendinopathy with symptoms present ≥8 weeks but <12 months at screening.
* The Achilles tendinopathy must have been refractory to at least 6 weeks of conservative treatment (physiotherapy, NSAIDS, RICE), but participants do not need to be in physiotherapy at the time of study entry.

Exclusion Criteria:

* Medical condition that would affect safety of peritendon injection (e.g., peripheral vascular disease, use of anticoagulant medication)
* History of recurrent, acute, symptomatic infections, including outbreaks of oral or genital herpes (> 2 symptomatic infections or >2 courses of anti-infective treatments required in the last 6 months; active systemic infection during last 2 weeks; known active infections (e.g. chronic or active Hepatis B or C, HIV) - simple cold excluded
* History or evidence of clinically significant cardiac or cardiovascular disease
* History of deep vein thrombosis, pulmonary embolism or evidence of primary or secondary hypercoagulable states
* History of surgical intervention for the treatment of tendinopathy, history of ankle surgery, ankle arthritis, traumatic, inflammation or deformity of ankle
* History of full-thickness tear or complete rupture of the Achilles tendon

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with AEs and SAEs | Up to Day 169 (End of Study)
  AEs and SAEs including ECG parameters, Lab Chemistry and Hematology parameters, urinalysis, local tolerability

SECONDARY OUTCOMES:
Changes in tendon stiffness from baseline at week 12 assessed by ultrasound (US)-based shear wave elastography (SWE) | Baseline, Week 12
  To assess the effects of a single peritendon injection of NGI226 MP versus placebo on restoration of biomechanical integrity of Achilles tendon

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Tucson Orthopedic Institute PC, Tucson, Arizona
  - Advanced Research LLC, Deerfield Beach, Florida
  - Houston Methodist Hospital, Houston, Texas
- Novartis Investigative Site, Caluire-et-Cuire, France
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided